CLINICAL TRIAL: NCT05463172
Title: Comparison Of Abdominal Muscles Strengthening And Pelvic Floor Muscle Strengthening Exercises On Bladder Neck Mobility In Females With Urinary Incontinence
Brief Title: Abdominal Muscles Strengthening And Pelvic Floor Muscle Strengthening Exercises In Females With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0526
Record Dates: First submitted 2022-04-15; First posted 2022-07-18 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Urinary Incontinence
Keywords: bladder neck mobility
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor muscles strengthening exercises (Experimental): pelvic floor muscles strengthening exercises
  Interventions: Other: pelvic floor muscles strengthening exercises
- abdominal strengthening exercises (Experimental): abdominal strengthening exercises
  Interventions: Other: abdominal strengthening exercises

INTERVENTIONS:
Other: abdominal strengthening exercises — abdominal strengthening exercises
  Arms: abdominal strengthening exercises
Other: pelvic floor muscles strengthening exercises — to strengthen pelvic floor muscles
  Arms: pelvic floor muscles strengthening exercises

SUMMARY:
Urinary incontinence is common females., it badly affects their performance and result in psychosocial problems in addition to the barriers that already have been resulted from incontinence. This study combines simple regime of hip adductor a strengthening with pelvic floor muscles. The theme is to test if pelvic floor muscle training can be augmented by incorporating adductor muscle strengthening. If this comes out to be effective, this can be great contribution to gym doing females to improve their urinary incontinence related impairments. Woman would be encouraged to continue regular exercise. This will be randomized clinical trial. There are two groups for the compression of adductors strengthening and pelvic floor muscle strengthening.

The collected data will be entered in SPSS 20.0, Descriptive and Inferential statists will be applied. Results and conclusion will be drawn.

DETAILED DESCRIPTION:
Urinary incontinence is common females., it badly affects their performance and result in psychosocial problems in addition to the barriers that already have been resulted from incontinence. This study combines simple regime of hip adductor a strengthening with pelvic floor muscles. The theme is to test if pelvic floor muscle training can be augmented by incorporating adductor muscle strengthening. If this comes out to be effective, this can be great contribution to gym doing females to improve their urinary incontinence related impairments. Woman would be encouraged to continue regular exercise. This will be randomized clinical trial. There are two groups for the compression of adductors strengthening and pelvic floor muscle strengthening.

Group A: with pelvic floor muscle strengthening is strengthening. Group B: abdominal muscles strengthening exercises. The collected data will be entered in SPSS 20.0, Descriptive and Inferential statists will be applied. Results and conclusion will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-45 years of age
* Females with abdominal muscles weakness
* Females with pelvic floor muscles weakness
* Females with urinary incontinence

Exclusion Criteria:

* Pregnant females
* Females having any history of trauma
* Any neurological disorders affecting bowl bladder
* Any malignancy in lower abdominal area

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female only
Enrollment: 22 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
urinary distress | 6 months
  Urinary Distress Inventory, Short Form (UDI-6), UDI-6 consists of 6 items: 1-Frequent urination, 2-Leakage related to feeling of urgency, 3-Leakage related to activity, 4-Coughing, or sneezing small amounts of leakage (drops), 5-Difficulty emptying the bladder, and 6-Pain or discomfort in the lower abdominal or genital area
Cough stress test | 6 months
  Cough stress test to evaluate urinary incontinence. Leakage of fluid from the urethral meatus coincident with/simultaneous to the cough(s) is considered a positive test.
Vaginal Ultrasonography | 6 months
  Bladder neck mobility can be described as a semicircular movement with the tip of the symphysis pubis as the center and a line from the tip to the bladder neck as the radius (BS). Movement can be measured by 2 independent factors: BS distance and size of the angle between the BS line and the midline of the symphysis, at rest, during the Valsalva maneuver and withholding urine. The continent controls were characterized by a 90 degrees angle at rest, a long BS (2.4 cm) and a fixed bladder neck

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Jinah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneeweiss J, Koch M, Umek W. The human urinary microbiome and how it relates to urogynecology. Int Urogynecol J. 2016 Sep;27(9):1307-12. doi: 10.1007/s00192-016-2944-5. Epub 2016 Jan 25. PMID 26811114
- [Background] Al-Mukhtar Othman J, Akervall S, Milsom I, Gyhagen M. Urinary incontinence in nulliparous women aged 25-64 years: a national survey. Am J Obstet Gynecol. 2017 Feb;216(2):149.e1-149.e11. doi: 10.1016/j.ajog.2016.09.104. Epub 2016 Oct 6. PMID 27720862
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322